CLINICAL TRIAL: NCT00810602
Title: Phase II Trial of Vorinostat Plus Tacrolimus & Mycophenolate to Prevent Graft Versus Host Disease Following Reduced Intensity Conditioning Related Donor Allogeneic Transplant
Brief Title: Vorinostat to Prevent Graft Versus Host Disease Following Reduced Intensity, Related Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pavan Reddy, MD (Other)
Responsible Party: Sponsor-Investigator, Pavan Reddy, MD, Professor, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2008.095
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Hematologic Malignancies; Graft vs Host Disease
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — Tacrolimus; Mycophenolic Acid; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat prophylaxis (Experimental): Vorinostat,combined with standard GVHD prevention medications(tacrolimus, mycophenolate) for adults who received a reduced intensity, related donor stem cell transplant
  Interventions: Procedure: reduced intensity, related donor stem cell transplant; Drug: tacrolimus (standard GVHD prophylaxis); Drug: mycophenolate (standard GVHD prophylaxis); Drug: vorinostat

INTERVENTIONS:
Procedure: reduced intensity, related donor stem cell transplant — Fludarabine /Busulfan(FluBu2)regimen
  Fludarabine: 40 mg/m2/day in 0.9 NS, administered IV on days -5 to day -2 pre-transplant for a total of 4 doses. Busulfan: 3.2 mg/kg in 0.9 NS administered IV on days -5 and -4 for a total of 2 doses. Total body irradiation 200 cGy delivered in a single fraction will be given on day 0 for patients receiving an HLA-mismatched transplant.
Drug: tacrolimus (standard GVHD prophylaxis) — Tacrolimus will begin on day -3, IV or oral. Target trough level for tacrolimus is 8-12 ng/ml. In the absence of GVHD, tacrolimus tapering will begin on day +56 post transplant
Drug: mycophenolate (standard GVHD prophylaxis) — Mycophenolate will begin on day 0 at 10 mg/kg/dose (up to 1 gram per dose) every 8 hours orally or intravenously and will continue until day 28.
Drug: vorinostat — Vorinostat given at a dose 100 mg PO BID starting day -10. If tolerated, vorinostat will be continued until day 100 post-transplant,whether or not acute GVHD develops.
  Dose escalation/ de-escalation
  Ten subjects treated at a dose of 100 mg PO BID. If dosing modifications are not required, during the pre-engraftment period in more than 4 patients, AND no more than two observed drug related toxicities CTC grade 4 or higher [probably or definitely related to the drug] then vorinostat dose will be escalated to 200 mg PO BID.
  If dose escalation does not occur due to failure to meet the above criteria,then the study will enroll at the 100 mg PO BID dosing, subject to the protocol stopping rules.
  If dose escalation occurs, subjects will be treated at 200 mg PO BID dosing level. If the probability of unacceptable toxicity exceeds the rules in protocol, then the dose of vorinostat will be de-escalated to 100 mg PO BID for the remainder of study.
  Other Names: ZOLINZA

SUMMARY:
The proposed research study is to test the drug vorinostat, in a new use as an additional medication, with other standard treatments for the prevention of severe acute graft versus host disease (GVHD).

If this treatment is safe and effective, when combined with a reduced intensity transplant, the research may achieve a more effective therapy for patients with high-risk, blood cell related cancers.

All subjects will receive an identical, known treatment to test if the treatment is safe and effective (a phase II trial). For patients to take part they must have a high-risk, blood cell cancer, be suitable candidates to receive a reduced intensity transplant and have a matched, related donor.

Adult subjects (age 18 years and older) will be considered as subjects provided, as detailed in the protocol, they meet additional criteria and are not excluded from participating. About fifty (50) subjects will be enrolled in this study at the University of Michigan.

Patients who receive blood stem cell transplants (HSCT), also called bone marrow transplants, to treat their cancer are at risk for serious complications, which may sometimes be fatal. The more common, serious ones are relapse (return of their disease), body organ injury from the intensity of the chemotherapy given prior to their transplant, and a serious complication called graft versus host disease (GVHD). GVHD is a form of rejection, where the transplanted cells of the donor attack the recipient's body as foreign, and do damage to organs and tissues.

To decrease the side effects of the chemotherapy given before a transplant, reduced intensity treatment plans(regimens)have recently been developed at a number of transplant centers. A decrease in the side effects of chemotherapy (called toxicities) has been achieved; however, this success with "less intensive" treatments has been partially offset by less successful results in controlling the patient's cancer.

As mentioned above, GVHD is a form of transplant rejection. GVHD can affect the digestive system, skin, liver and other body systems. GVHD can increase the risk of infection. After a matched, related donor stem cell transplant, GVHD when severe, is a major cause of discomfort, organ damage, and even death. When a graft vs host reaction develops, but is kept under control, studies show there may be a beneficial graft versus tumor effect, helping to destroy tumor cells in the patient, and thus providing a more effective control of their cancer.

The goal of this study is to try to maximize the potential benefits, of giving patients less intense chemotherapy to reduce the toxic effects, letting the graft vs host effect help in destroying tumor cells, but preventing acute severe GVHD by using the drug vorinostat, combined with standard medicines, to reduce the chance of serious GVHD-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Have a 7/8 or 8/8 HLA A, B, C and DR, HLA-matched related donor willing and able to donate allogeneic stem cells.
* For patients with multiple myeloma, CLL, and lymphoma: must be in CR, PR, or stable disease.
* For MDS, acute leukemia or CML: must have <20% blasts on marrow exam.
* For all other diseases: must have non-refractory disease.

and meet at least ONE of the next three criteria:

* Any patient ≥ 18 years of age with a hematological malignancy and not considered a candidate for allogeneic myeloablative transplant due to illness and/or age (≥55 years).
* Any patient ≥ 18 years of age who has relapsed following prior autologous or allogeneic transplant for a hematologic malignancy.
* Any patient ≥ 18 years of age diagnosed with a hematological malignancy for which reduced intensity transplant is institutionally preferred over myeloablative transplant (eg, chronic lymphocytic leukemia).

Exclusion Criteria:

* Less than 18 years of age.
* Currently taking any HDAC inhibitors, or have taken an HDAC inhibitor within 30 days of the trial.
* Positive serum tests for HIV, HTLV1 / HTLV2.
* Detectable hepatitis B virus (HBV), hepatitis C (HCV) or Epstein-Barr (EBV).
* Pregnancy.
* One or more of the following organ system function criteria

  * Cardiac: Ejection fraction ≤ 40%
  * Renal: Estimated or actual GFR ≤ 40 ml/min (corrected for BSA)
  * Pulmonary: FEV1, FVC, or DLCO ≤ 40% predicted
  * Hepatic: Total bilirubin ≥3 mg% and AST/ALT >5 x institutional normal for age
  * Karnofsky score ≤50 (Requires considerable assistance and frequent medical care).
* Persistent invasive infections not controlled by antimicrobial medication.
* Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Reddy, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Result] Choi SW, Braun T, Chang L, Ferrara JL, Pawarode A, Magenau JM, Hou G, Beumer JH, Levine JE, Goldstein S, Couriel DR, Stockerl-Goldstein K, Krijanovski OI, Kitko C, Yanik GA, Lehmann MH, Tawara I, Sun Y, Paczesny S, Mapara MY, Dinarello CA, DiPersio JF, Reddy P. Vorinostat plus tacrolimus and mycophenolate to prevent graft-versus-host disease after related-donor reduced-intensity conditioning allogeneic haemopoietic stem-cell transplantation: a phase 1/2 trial. Lancet Oncol. 2014 Jan;15(1):87-95. doi: 10.1016/S1470-2045(13)70512-6. Epub 2013 Nov 30. PMID 24295572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2008 through February 2013, eligible patients with advanced hematological cancers were enrolled at the University of Michigan and Washington University in St. Louis.
Pre-assignment Details: All patients received a preparative regimen of intravenous fludarabine (40 mg/m2 on day -5 through day -2) and busulfan (3.2 mg/kg on days -5 and -4) (FluBu2) followed by the infusion of peripheral blood stem cells (PBSC) on day 0. GVHD prophylaxis consisted of tacrolimus initiated on day -3 and mycophenolate mofetil (MMF) on day 0 through day 28.
Groups:
- Phase 1: In the Phase 1 portion of the study, participants were administered Vorinostat, either 100 mg or 200mg, twice daily, orally, starting ten days prior to the stem cell infusion and continuing through day 100 post-HSCT. If tolerated, vorinostat will be continued until day 100 post-transplant,whether or not acute GVHD develops.
- Phase 2: 100 mg was selected as the Phase 2 dose. Participants were administered Vorinostat, 100 mg, twice daily, orally, starting ten days prior to the stem cell infusion and continuing through day 100 post-HSCT. If tolerated, vorinostat will be continued until day 100 post-transplant,whether or not acute GVHD develops.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 27 | 34
Completed | 19 | 31
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Population: Only participants that completed 21 days of vorinostat were considered evaluable for both toxicity and the primary outcome, therfore only 50 of the 61 patients initially enrolled are represented in baseline characteristics.
Groups:
- Vorinostat Prophylaxis: Vorinostat, combined with standard GVHD prevention medications(tacrolimus, mycophenolate) for adults who received a reduced intensity, related donor stem cell transplant.
  Vorinostat was administered daily starting ten days prior to the stem cell infusion and continued through day 100 post-HSCT. If tolerated, vorinostat will be continued until day 100 post-transplant,whether or not acute GVHD develops.
  The phase 1 portion of the study tested two doses of vorinostat, 100 mg BID and 200 mg BID.The first ten patients received vorinostat 100 mg BID, followed by nine patients who received the 200 mg BID dose.
  Although no dose-limiting toxicities were reached at the 200 mg BID dose, there was an increased incidence of protocol-driven dose modifications, primarily due to non-symptomatic thrombocytopenia after engraftment. Consequently, the 100 mg BID dose was selected as the phase 2 dose for the remaining patients.
Arm/Group | Vorinostat Prophylaxis
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — (44%, 56% of evaluable subjects, respectively)
  Participants
    Female | 22
    Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Diagnosis [Number; unit: participants]
  Acute myelogenous leukemia | 19
  Myelodysplastic syndrome | 10
  Non-Hodgkin's lymphoma | 12
  Chronic lymphocytic leukemia | 4
  Myeloproliferative disorder or myelofibrosis | 4
  Acute biphenotypic leukemia | 1
Disease Status [Number; unit: participants]
  Low | 25
  Intermediate | 20
  High | 5
Comorbidity index [Number; unit: participants] — Hematopoietic Cell Transplant - Comorbidity Index: Low = 0, Intermediate = 1 or 2, High ≥ 3
  participants
    Low | 8
    Intermediate | 15
    High | 27
Donor Type [Number; unit: participants]
  Matched related | 46
  One-antigen mismatched related | 4
CMV Status [Number; unit: participants] — Recipient(R),Donor (D), positive (+), negative(-)
  participants
    Recipient or Donor positive (detailed below) | 30
    R+, D+ | 17
    R-, D+ | 6
    R+, D- | 7
    Recipient and Donor negative | 20
CD34+ Count (10^6 cells/kg) [Median (Full Range); unit: Count (10^6 cells/kg)] | 5.0 [1.9 to 8]
Engraftment Day [Median (Full Range); unit: days] — Median time to platelet and neutrophil engraftment.
  days
    Neutrophil | 12 [8 to 19]
    Platelet | 12 [9 to 30]

OUTCOME MEASURES:

1. Primary Outcome: 100-day Cumulative Incidence of Grade 2-4 Acute Graft Versus Host Disease (GVHD)
Description: Assess if the addition of Vorinostat to standard GVHD prophylaxis regimen can reduce the rate of grades 2-4 acute GVHD when compared to 48% in a cohort of identically treated RIC HSCT patients without vorinostat. A reduction of incidence to less than 25% will be considered successful.
Time Frame: 100 days
Population: evaluable
Measure: Number; unit: percentage of participants
Groups:
- Vorinostat Prophylaxis: Vorinostat,combined with standard GVHD prevention medications(tacrolimus, mycophenolate) for adults who received a reduced intensity, related donor stem cell transplant.
  Vorinostat was administered daily starting ten days prior to the stem cell infusion and continued through day 100 post-HSCT. If tolerated, vorinostat will be continued until day 100 post-transplant,whether or not acute GVHD develops.
  The phase 1 portion of the study tested two doses of vorinostat, 100 mg BID and 200 mg BID.The first ten patients received vorinostat 100 mg BID, followed by nine patients who received the 200 mg BID dose.
  Although no dose-limiting toxicities were reached at the 200 mg BID dose, there was an increased incidence of protocol-driven dose modifications, primarily due to non-symptomatic thrombocytopenia after engraftment. Consequently, the 100 mg BID dose was selected as the phase 2 dose for the remaining patients.
Arm/Group | Vorinostat Prophylaxis
Number analyzed (Participants) | 50
percentage of participants | 22
Statistical Analysis 1: Comparison: Vorinostat Prophylaxis; Hypothesis: The addition of vorinostat will reduce the incidence of grade 2-4 acute graft versus host disease (GVHD) to 25% or lower by day 100; Test type: Superiority or Other; Percent Cumulative Incidence of GVHD = 22, 95% CI 2-sided [13 to 36]

2. Secondary Outcome: Number of Serious Adverse Events
Description: The safety and feasibility will be partially measured by the number of serious adverse events (SAE) recorded by participants receiving at least one dose of Vorinostat.
Time Frame: 100 days
Population: The number of patients who received at least one dose of vorinostat.
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Vorinostat Prophylaxis
Number analyzed (Participants) | 58
Number of Serious Adverse Events | 33

3. Secondary Outcome: Percent Cumulative Incidence of Relapse at 2 Years.
Description: Determine the cumulative incidence of relapse at 2 years.
Time Frame: two years
Population: evaluable subjects
Measure: Number; unit: percentage of participants
Arm/Group | Vorinostat Prophylaxis
Number analyzed (Participants) | 50
percentage of participants | 16
Statistical Analysis 1: Comparison: Vorinostat Prophylaxis; Test type: Superiority or Other; Percent Cumulative Incidence of GVHD = 16, 95% CI 2-sided [8 to 30]

4. Secondary Outcome: Percent Survival at 2-years
Description: To determine 2-year overall survival rate
Time Frame: two years
Population: evaluable subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Vorinostat Prophylaxis
Number analyzed (Participants) | 50
percentage of subjects | 73

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from March 2008 through April of 2013.
Arm/Group | Vorinostat Prophylaxis
Serious Adverse Events (participants affected / at risk) | 31/58
Other Adverse Events (participants affected / at risk) | 51/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat Prophylaxis (N=58)
Anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Edema: Limb (General disorders) | 1
Hemmorrhoids (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 12
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Graft Versus Host Disease (Immune system disorders) | 5
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat Prophylaxis (N=58)
Alanine Aminotransferase Increased (Investigations) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 29 (45)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Infection (Infections and infestations) | 8 (8)
Leukocytes (White Blood Cells Decreased) (Investigations) | 51 (84)
Lymphopenia (Investigations) | 50 (109)
Neutrophils Decreased (Investigations) | 50 (100)
Platelets Decreased (Investigations) | 50 (184)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes